# **COVER PAGE**

## Official Title of the Study:

Comparative Effects of BCI-Based Attention Training, Methylphenidate, and Citicoline on Attention and Executive Function in School-Age Children: A Naturalistic Quasi-Experimental Study

## **ClinicalTrials.gov Identifier (NCT Number):**

"Not yet assigned"

## **Document Type:**

Informed Consent Form (Parental Permission Form)

#### **Document Date:**

16 December 2025

### **INFORMED CONSENT FORM (Parental Permission Form)**

**Study Title:** Comparative Effects of BCI-Based Attention Training, Methylphenidate, and Citicoline on Attention and Executive Function in School-Age Children: A Naturalistic Quasi-Experimental Study

**Principal Investigator**: Assoc. Prof. Serkan Turan, MD Department of Child and Adolescent Psychiatry Bursa Uludağ University Faculty of Medicine, Turkey

#### Introduction

Your child is invited to participate in a research study because of attention-related difficulties. Participation is voluntary, and you may withdraw your child at any time without affecting care.

#### Purpose of the Study

The purpose of this study is to compare different clinical approaches used to support attention and executive functioning in school-aged children.

### **Study Procedures**

Your child will complete routine clinical assessments, computerized attention tasks, and may receive BCI-based attention training, medication, citicoline, or combinations as part of standard care.

### Duration

Participation will last approximately 8 weeks.

## **Risks and Discomforts**

This study involves minimal risk, similar to routine clinical practice.

## **Potential Benefits**

Your child may or may not directly benefit. The study may help improve future treatments. Confidentiality All data will be kept confidential and de-identified.

# **Voluntary Participation**

You may withdraw your child at any time without penalty.

## **Contact Information**

Assoc. Prof. Serkan Turan, MD Email: <a href="mailto:serkanturan@uludag.edu.tr">serkanturan@uludag.edu.tr</a>

#### **Statement of Consent**

I have read and understood the information above and voluntarily agree to my child's participation.

| Parent/Guardian Name: _ | <br> |
|-------------------------|------|
| Signature: | |
| Date: | |